CLINICAL TRIAL: NCT00920725
Title: Subcutaneous Aspart Insulin and Point of Care Beta Hydroxybutyrate Testing: A New Paradigm for the Management of Diabetic Ketoacidosis
Brief Title: Subcutaneous Aspart Insulin to Treat Diabetic Ketoacidosis (DKA) and Beta-Hydroxybutyrate Testing in DKA
Acronym: DKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, David Baldwin, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05012103
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Diabetic Ketoacidosis
Keywords: DKA
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Subcutaneous Insulin (Active Comparator): Aspart Insulin administered subcutaneously 0.2 units/kg/sq every 2 hours
  Interventions: Drug: Insulin (Aspart Insulin [Novolog], Regular Insulin)
- IV Regular Insulin (Active Comparator): Intravenous Regular Insulin 0.1 units/kg/hour
  Interventions: Drug: Insulin (Aspart Insulin [Novolog], Regular Insulin)
- Intravenous Novolog Insulin (Active Comparator): Intravenous Novolog Insulin 0.1 units/kg/hour
  Interventions: Drug: Insulin (Aspart Insulin [Novolog], Regular Insulin)

INTERVENTIONS:
Drug: Insulin (Aspart Insulin [Novolog], Regular Insulin) — Aspart Insulin 0.2units/sq q 2 hours
  Regular Insulin 0.1units/kg/hr intravenous
  Aspart Insulin 0.1 units/kg/hr intravenous

SUMMARY:
The purpose of this study is to determine whether insulin administered by a subcutaneous injection is effective in the treatment of a diabetic crisis and to determine if beta-hydroxybutyrate is useful to monitor during treatment of a diabetic crisis.

ELIGIBILITY:
Inclusion Criteria: age 18 or older

* venous pH < 7.3 or arterial < 7.35
* at least 2 of the following 3:

  1. serum HCO3 < 18/anion gap > 16
  2. serum glucose > 300 mg/dl
  3. serum acetone positive

Exclusion Criteria:

* pregnant
* less than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hours to resolution of ketoacidosis as defined as beta-hydroxybutyrate <0.6 | q 2 hours
Hours to achieve blood glucose less than 200mg/dl | q 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Rema A Gupta, MD, Principal Investigator — Rush University Medical Center; David Baldwin, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States